CLINICAL TRIAL: NCT06523959
Title: Avoiding Risks of Thrombosis and Bleeding in Surgery (ARTS) Trial: An International Randomised Controlled Trial Evaluating Apixaban Versus No Anticoagulation in Patients Undergoing General Abdominal, Gynecologic and Urologic Surgery
Brief Title: Avoiding Risks of Thrombosis and Bleeding in Surgery (ARTS) Trial
Acronym: ARTS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Urology and Epidemiology Working Group (Other Government)
Collaborators: Helsinki University Central Hospital (Other); University of Helsinki (Other); University College, London (Other); Population Health Research Institute (Other); Tabriz University of Medical Sciences (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); North Karelia Central Hospital (Other); Albany Medical College (Other); PaijatHame Central Hospital (Other)
Responsible Party: Principal Investigator, Kari Tikkinen, Professor of Urology, University of Helsinki and Helsinki University Hospital, Clinical Urology and Epidemiology Working Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLUE-ARTS-2023; 2023-508147-43-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-05; First posted 2024-07-29 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Venous Thromboembolism; Bleeding
Keywords: angioembolisation; apixaban; bleeding; complications; deep vein thrombosis; direct oral anticoagulant; DOAC; embolisation; evidence-based medicine; gynecology; hemoglobin; hemorrhage; mortality; open label; postoperative; pragmatic; pulmonary embolism; randomized trial; RCT; re-operation; reintervention; surgery; thrombosis; thromboprophylaxis; transfusion; urology; venous thromboembolism; VTE
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage; Venous Thrombosis; Pulmonary Embolism; Thrombosis | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: This is a pragmatic randomized controlled, parallel group, open-label trial with a 1:1 randomization (block randomization) ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apixaban (Experimental): Apixaban 2.5mg (i.e Eliquis® 2,5mg tablet) orally twice daily for 28 days (with standard of care mechanical prophylaxis)
  Interventions: Drug: Apixaban 2.5 MG
- No anticoagulation (No Intervention): No anticoagulation (with standard of care mechanical prophylaxis)

INTERVENTIONS:
Drug: Apixaban 2.5 MG — To evaluate the benefits and risks of thromboprophylaxis with oral factor Xa inhibitor Apixaban compared to No anticoagulation
  Other Names: Eliquis 2,5mg
  Arms: Apixaban

SUMMARY:
Avoiding Risks of Thrombosis and bleeding in Surgery (ARTS) trial is a pragmatic, international, multicenter, randomized controlled open label trial comparing a direct oral anticoagulant (DOAC) - oral factor Xa inhibitor apixaban - to no anticoagulant among 5,436 patients undergoing abdominal or pelvic surgery at sufficiently similar (and not high) risk of venous thromboembolism (VTE) and bleeding that the net impact - benefit or harm - of thromboprophylaxis remains in doubt.

DETAILED DESCRIPTION:
Deep vein thrombosis and pulmonary embolism - collectively known as venous thromboembolism VTE - and major bleeding are serious surgical complications leading to poorer patient-reported quality of life and mortality. Pharmacological thromboprophylaxis is an established strategy for reducing VTE risk but balancing it with increased bleeding, particularly after major surgery, poses challenges. Guidelines typically recommend pharmacological thromboprophylaxis for patients at higher, but not lower risk of VTE, without clearly defining procedure or patient selection. There is particular uncertainty regarding the balance of potential benefits and harms of pharmacological thromboprophylaxis in patients who are at a lower estimated risk of VTE postoperatively, in patients with a baseline VTE risk in the range of 2%. In these patients, the risk of major bleeding may be similar to or could potentially outweigh the relatively lower risk of VTE complications, such that the net clinical benefit of routine pharmacological thromboprophylaxis remains unclear.

"Avoiding Risks of Thrombosis and Bleeding in Surgery (ARTS)" is a large, randomized, multicenter study, comparing a direct oral anticoagulant (DOAC) called apixaban in patients undergoing abdominal and pelvic surgeries. Half of the 5436 patients will be randomized to receive apixaban after surgery for 28 days with standard of care mechanical prophylaxis - to a control group with no anticoagulation but with standard of care mechanical prophylaxis.

ARTS trial will be the first to compare anticoagulation with DOACs (apixaban) versus no anticoagulation in a population of urologic, gynecologic and abdominal surgical patients. Any of the possible outcomes of 1) A clear net benefit in favor of apixaban or 2) A clear net benefit to not using prophylaxis or 3) a sufficiently close tradeoff that predictive factors and patients' values and preferences regarding bleeding versus thrombosis determines the decision, will substantially enhance evidence-based peri-operative care.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided
* Adult patients (≥18 years);
* Undergoing elective abdominal or pelvic surgery at similar (and not high) risk of VTE and bleeding

Exclusion Criteria:

* Inability to provide informed consent
* Patient with active bleeding/hemorrhage during the last 6 months if not expected to be treated by surgery planned
* Lesion or condition if considered a significant risk factor for major bleeding

  a. This may include current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities
* Anticoagulant treatment, antiplatelet treatment or omega-3 dietary supplement during previous 7 days preceding surgery and/or requiring within 30 days post-surgery
* Patient who had during previous 6 months or are expected require within 30 days post-surgery chemotherapy/radiation or hormone therapy for cancer
* Known thrombophilia
* Known bleeding disorder
* Substantial liver impairment (for instance INR 1.4 or more during last 60 days)
* eGRF <30 mL/min/1.73 m2
* Platelet count <100 × 109/L (that is, 100 000 mg/L)
* Hb <90 g/L (that is, <9 g/dL)
* ALT >2 × upper limit of normal
* Known allergy to apixaban
* Taking strong inhibitors or inductors of both CYP 3A4 and P-glycoprotein, such as anti-seizure medications (e.g. phenytoin, fosphenytoin, carbamazepine), azole-antimycotics (e.g. ketoconazole, itraconazole), HIV-protease inhibitors (e.g. ritonavir, indinavir) and rifampicin
* Concomitant procedures with high risk of VTE/bleeding
* Previous VTE
* Pregnant or breast-feeding female patients
* Female participants who have had periods in the last 12 months and who are not using highly reliable contraception: (i) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); ii) progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); iii) intrauterine device (IUD); iv) intrauterine hormone-releasing system (IUS); v) bilateral tubal occlusion; vi) vasectomized partner; and vii) sexual abstinence from heterosexual intercourse during the entire period of risk associated with the study treatments
* Previous randomization in this trial
* Any reason why, in the opinion of the investigator(s), the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5436 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence composite outcome of venous thromboembolism (VTE) | 90 days
  Defined as symptomatic deep vein thrombosis (DVT), or symptomatic non-fatal or fatal pulmonary embolism (PE)

SECONDARY OUTCOMES:
Incidence of symptomatic DVT | 90 days
  Defined as symptomatic deep vein thrombosis
Incidence of symptomatic PE | 90 days
  Defined as symptomatic non-fatal of fatal pulmonary embolism (PE)

OTHER OUTCOMES:
Incidence of composite endpoint for major bleeding | 90 days
  Defined as composite endpoint of bleeding leading to a postoperative hemoglobin <70 g/L, transfusion of ≥1 unit of red blood cells, or bleeding that was judged to be the immediate cause of death
Incidence of re-intervention or endovascular embolization to stop bleeding | 90 days
  Defined as bleeding requiring re-intervention or endovascular embolization to stop bleeding
Incidence of composite outcome of VTE | 30 days
  Defined as symptomatic DVT, or symptomatic non-fatal or fatal PE
Incidence of composite endpoint for major bleeding | 30 days
  Defined as composite endpoint of bleeding leading to a postoperative hemoglobin <70 g/L, transfusion of ≥1 unit of red blood cells, or bleeding that was judged to be the immediate cause of death
Incidence of re-intervention or endovascular embolization to stop bleeding | 30 days
  Defined as bleeding requiring re-intervention or endovascular embolization to stop bleeding
Incidence of symptomatic non-fatal PE | 90 days
  Defined as symptomatic non-fatal pulmonary embolism
Incidence of symptomatic fatal PE | 90 days
  Defined as fatal pulmonary embolism
Incidence of bleeding leading to a postoperative hemoglobin <70 g/L | 90 days
Incidence of transfusion of ≥1 unit of red blood cells | 90 days
Incidence of bleeding that was judged to be the immediate cause of death | 90 days
Incidence of bleeding requiring re-intervention to stop bleeding | 90 days
Incidence of bleeding requiring endovascular embolization to stop bleeding | 90 days
Overall mortality | 90 days
Incidence of SUSARs potentially related to the study drug (apixaban) | 90 days
Incidence of Serious Adverse Events (SAEs), any | 90 days
Incidence of any potentially drug-related SAEs (serious), cardiac complications, cerebral complications, infectious complications, admittance to intensive care, reoperation or other intervention for other reason than bleeding and other complication | 90 days
Incidence of critical organ bleeding | 90 days
Cost-effectiveness of DOAC administration | 90 days
  The trial will also assess the cost-effectiveness of apixaban administration compared to no pharmacological thromboprophylaxis. An extended time horizon decision analytic model will evaluate the costs associated with VTE and bleeding events in both trial arms. Based on these analyses, the additional or saved costs per quality- adjusted life-year (QALY) will be determined for various trial outcomes, including scenarios where apixaban is superior to no pharmacological thromboprophylaxis or vice versa. Costs will be evaluated from the perspective of national health service in selected countries. This assessment will consider patient healthcare resource utilisation, staff training costs (e.g., administering subcutaneous injections), and medication costs. The benefits of the interventions will be measured in terms of clinical outcomes, such as the reduction in VTE events and complications (including VTE and bleeding events). Additionally, QoL information will be used to calculate QALYs.

CONTACTS AND LOCATIONS:
Overall Officials: Kari AO Tikkinen, Professor, Principal Investigator — University of Helsinki and Helsinki University Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
The research data needed to validate the results presented in the deposited scientific publications are deposited and the data of individual participants is made available to the research community. Incase the publication would mean disclosing information relating to the Party's Confidential Information the Parties shall negotiate how to modify the publication in order to remove such Confidential Information from the publication. In case the publication would prevent a Party from securing its Intellectual Property Rights the publication shall be postponed until the rights have been secured.
Time Frame: Not longer than sixty (60) days from the claim made to restrict the publication.
Access Criteria: If the Parties have not expressed their well-founded and specified claim to restrict the publication within the said time limit, the publication shall be considered permitted.